CLINICAL TRIAL: NCT06291584
Title: Effects of Strengthening and Respiratory Exercises on Face and Online on Functional Capacity
Brief Title: Effects of Exercises on Functional Capacity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Fulya Demirhan, Research Assistant, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20230001
Record Dates: First submitted 2024-02-09; First posted 2024-03-04 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Nicotine Addiction; Respiratory Disease; Sedentary Behavior
Keywords: nicotine addiction; respiratory exercise; telehealth; resistance exercise
MeSH Terms: conditions — Tobacco Use Disorder; Respiration Disorders; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study consists of three groups. Groups to be formed: Group 1: face-to-face exercise group; Group 2: Online (Telehealth) Exercise Group; Group 3: Control Group
Who Masked: Participant
Masking Description: First of all, the randomization of exercise groups will be performed according to the closed envelope procedure. The student who selects one of the envelopes with the names of the three groups will be included in the group written in the envelope he selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-Face Exercise Group (Experimental): In the face-to-face exercise group called Group 1, students will apply an exercise program of respiratory exercises and resistance exercises with the physiotherapist.
  Interventions: Other: Exercise
- Telehealth Exercise Group (Experimental): In the online (telehealth) exercise group, group 2 will be applied by the students with the help of the physiotherapist.
  Interventions: Other: Exercise
- Control Group (No Intervention): In the control group called Group 3, students will not be given any exercise program.

INTERVENTIONS:
Other: Exercise — In the exercise program, the first 5 minutes are for heating, and the last 5 minutes are for cooling. In the exercise program, which is planned to last 40 minutes in total, respiratory exercises will be applied to heating and cooling peryotes. At the end of respiratory exercises, resistance exercise training will be started. Elastic resistant bands (Therand) will be used in resistant exercise training that will last for 30 minutes. The participants will be started to work with the resistance that they can do 10 again but cannot reach 14 repetitions. Elastic resistant bands are shoulder flexion, shoulder extension, shoulder ablution, shoulder horizontal abduction, elbow extension, hip ablution, hip flexion, hip extrudy, squat, and cat-decrease. These exercises will be held once a week, 10 repetitions, 2 sets, for 8 weeks.
  Arms: Face-to-Face Exercise Group; Telehealth Exercise Group

SUMMARY:
In this study, the researchers aim to investigate the effects of strengthening and respiratory exercises on the face and online on functional capacity.

DETAILED DESCRIPTION:
The American Sports Medical Association has reported that a regular exercise program containing endurarans, strength, flexibility, and neuromotor exercise training is required in addition to daily life activities in order to maintain and develop general health. In addition to the increase in muscle strength with resistant exercises, durability and strength are also targeted. When performing resistant exercise, it is important to breathe correctly. The speed of the exercise and the movements are performed throughout the furnishing openness of the joint movement. The effects of exercise on being healthy and good are mentioned in the literature in detail. However, the effects of exercise on the respiratory functions and functional capacity of young people who smoke are not adequately defined. For this reason, the researchers plan to research the effects of strengthening and respiratory exercises on the face and online on functional capacity.

ELIGIBILITY:
Inclusion Criteria:

Signing the illuminated consent form, Being smoking at least 1 cigarette for the last 6 months, Not having orthopedic or neurological findings that can prevent the exercises included in the study, To have a low- to medium-level physical activity level, Not to have any lower respiratory infection in the last 3 months.

Exclusion Criteria:

The exercise sessions to be held on time and regularly.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | Evaluation should be carried out before the start of exercise proggramme and 8 weeks after.
  Validity and reliability work of the questionnaire in Turkey was conducted in 2010 by Sağlam and his friends. It has questions about the physical time spent in the last 7 days to learn about the physical activities of people in daily life.
Six-Minute Walk Test- (6MWT) | Evaluation should be carried out before the start of exercise proggramme and 8 weeks after.
  It is a widely used test for evaluating the functional capacity of individuals. Individuals are asked to walk at normal walking speeds for six minutes in a flat corridor of thirty meters long with a start and end point. The distance where cases walk for 6 minutes is recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu ÖZÜBERK, Assoc. prof., Principal Investigator — Kırklareli University
Locations (1):
- Kirklareli University, Kırklareli, Kayalı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided